CLINICAL TRIAL: NCT04969432
Title: Effectiveness of Client-centered Intervention Delivered With Face to Face and Telerehabilitation Method After Total Knee Arthroplasty - A Pilot Randomized Controlled Trial
Brief Title: Effectiveness of Client-centered Intervention in After Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Berkan Torpil, PhD, Principal Investigator, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Saglik Bilimleri Universitesi
Record Dates: First submitted 2021-07-08; First posted 2021-07-20 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Arthritis Knee
Keywords: Client-centered; Quality of life; Knee arthroplasty; Occupational performance; Telerehabilitation; Telemedicine
MeSH Terms: interventions — Person-Centered Psychotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation (Experimental)
  Interventions: Other: Client-centered
- Face-to-face (Experimental)
  Interventions: Other: Client-centered

INTERVENTIONS:
Other: Client-centered — Rehabilitation

SUMMARY:
The current study was conducted to comparison of the Client-centered (CC) intervention with face-to-face (FF) and TR methods after Total Knee Arthroplasty (TKA). The pilot study was planned to examine the impact of the CC intervention on quality of life, perceived occupational performance and satisfaction. The current study was designed according to the CONSORT statement, which provides a standardized method for randomized controlled trial (RCT) design. Approval for the study was granted by the Local Ethics Committee. Written informed consent was obtained from all participants prior to the study.

DETAILED DESCRIPTION:
The current study was conducted to comparison of the Client-centered (CC) intervention with face-to-face (FF) and TR methods after Total Knee Arthroplasty (TKA). The pilot study was planned to examine the impact of the CC intervention on quality of life, perceived occupational performance and satisfaction. The current study was designed according to the CONSORT statement, which provides a standardized method for randomized controlled trial (RCT) design. Approval for the study was granted by the Local Ethics Committee. Written informed consent was obtained from all participants prior to the study.

Participants A total of 56 older adults who were admitted to the occupational therapy department of a public university between January 2021 and May 2021 were screened. Participants who were eligible according to the evaluation and inclusion-exclusion criteria one week after TKA were included in the study. The study inclusion criteria were: (1) age between 65 and 75 years; (2) Mini Mental State Examination score of ≥24; (3) education level of at least completion of elementary school; (4) having undergone unilateral TKA surgery; (5) access to technological equipment; and (6) ability to understand and follow verbal instructions. The exclusion criteria were defined as: (1) revision surgery; (2) having any chronic disease that will affect the rehabilitation process; (3) auditory and visual problems that may affect rehabilitation implementation and communication; (4) postoperative complications (e.g., nerve injury and deep vein thrombosis); and (5) attendance of any rehabilitation program (physiotherapy, speech therapy, psychotherapy, etc.) during the study period.

Measurement The demographic characteristics of the participants were recorded, including age, sex, education level, body mass index (BMI), other people in the house where they lived, and marital status. The Mini Mental State Examination was used to determine the cognitive status included in the inclusion criteria. The Canadian Occupational Performance Measure and the Nottingham Health Profile were applied to all the subjects twice, before and after intervention.

Assessments Mini Mental State Examination Mini Mental State Examination (MMSE), which was used in the inclusion criteria of the study, was used to determine the cognitive state of the participants. From a maximum total of 30 points, a score of 24 is accepted as the threshold value, with scores below this value indicating problems in cognitive functions. Turkish validity and reliability studies of the test have been conducted and the researcher found the MMSE positive and negative predictive values .90 and .95 respectively and kappa score .86.

Canadian Occupational Performance Measure The Canadian Occupational Performance Measure (COPM) is a measure that determines the problems faced by individuals in the field of occupational performance through a semi-structured interview. Occupational performance problems are evaluated with self-reported performance and satisfaction scores. In the first step, ADL problems experienced by individuals in the areas of self-care, productivity and leisure are determined and each occupation is scored according to importance. The subject then selects a maximum of 5 occupations according to their importance scores and gives performance and satisfaction scores in a Likert-type system of 1- 10 for each occupation. The overall performance and satisfaction scores are obtained as the total of the performance and satisfaction scores of each occupation divided by the number of occupations. The Turkish version of COPM was used to evaluate the perceived occupational performance and satisfaction. The Turkish adaptation performed and test re-test reliability of Turkish version of COPM performance was .988 and satisfaction .986, indicating excellent reliability.

Nottingham Health Profile The Nottingham Health Profile (NHP) is a general quality of life questionnaire that measures perceived health problems and the level of these problems affecting normal ADL. The questionnaire consists of 38 items related to health status. Each item is answered as yes or no, and each section is scored between 0-100, with 0 indicating the best health status, and 100, the worst health status. In the Turkish adaptation study, test-retest reliability of the subscales (dimensions) of the scale varied between 0.70 and 0.92, and internal consistency values ranged between 0.56 and 0.87, confirming its validity and reliability.

Intervention The intervention program which was used both method (TR and FF) is designed to consist of 4 weeks, 4 days a week, 45-minute sessions. The caregiver actively participated in the treatment in order to prevent any possible injuries and to perform the applications more smoothly during the entire intervention process. The FF method was performed in the occupational therapy unit. The CC interventions with TR were delivered through real-time interaction programs such as Zoom, Skype, WhatsApp video call, or Microsoft Teams, according to the preference of the patient.

Client-centered intervention

The CC intervention developed according to the literature and based on a systematic therapy process, characterized by an active participatory attitude of both the participants after TKA process and the therapist, consisted of 5 phases: (1) CC goal-setting, (2) negotiating a therapy plan, (3) the actual intervention, (4) an evaluation of the outcome and (5) finally reporting to relevant others. The key aspect of this intervention was the CC approach in which the therapist is trained to clarify the prioritized goals of the patient. The therapy procedure was implemented according to the prioritized goals determined in the COPM. The stages are explained below:

First stage: Setting a measurable, realistic, and achievable goal for the solution of occupations involving performance problems.

Second stage: Develop and evaluate the pros and cons of possible solutions by brainstorming through the occupation determined with the COPM.

Third stage: After deciding on a possible solution, making a plan and taking action:

* Adaptation of the occupation determined with the COPM, making alterations to one or more of the following: who (involving another person), where (making a change in the place), when (changing the time), how (altering the way of application) and what (adding up new steps at the beginning or end of the occupation).
* Planning the steps of the occupation (in accordance with priority),
* Bringing together occupation-related information and resources

Fourth stage: Revising the therapy process which has been activated with the CC training

Fifth stage: Receiving feedback about individual's experiences and making alterations to the course of action when necessary.

Statistical analysis Data were analyzed with SPSS version 25.0 statistical software. Data were presented as mean ± standard deviation values. The conformity of the data to normal distribution was analyzed using the Kolmogorov-Smirnov test. The data were seen not to be distributed normally, so non-parametric statistical methods were used. Differences between groups were analyzed with the Chi-square test for nominal data. Comparisons between the groups were made using the Mann-Whitney U test. Pre- to post-intervention changes within the groups were analyzed with the Wilcoxon signed-rank test. Quade's rank analysis of covariance test was used to compare between group analysis. Statistical significance was evaluated at levels of 0.05.

The power of the study and effect sizes were analyzed using G*Power software, version 3.1.9.2. Power analysis was performed to calculate the sample size. It was determined that 21 subjects were needed in each group to ensure a power of 90%, assuming a two-tailed test for α equal to 0.05. Effect size was calculated using the means and standard deviations of the groups. Effect size benchmarks were determined as <0.30, 0.30-0.80, and >0.80, interpreted as small, moderate, and strong, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Age between 65 and 75 years
* Mini Mental State Examination score of ≥24
* Education level of at least completion of elementary school
* Having undergone unilateral TKA surgery
* Access to technological equipment
* Ability to understand and follow verbal instructions

Exclusion Criteria:

* Revision surgery
* Having any chronic disease that will affect the rehabilitation process
* Auditory and visual problems that may affect rehabilitation implementation and communication
* Postoperative complications (e.g., nerve injury and deep vein thrombosis)
* Attendance of any rehabilitation program (physiotherapy, speech therapy, psychotherapy, etc.) during the study period

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-01-07 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure | 40 minutes
Nottingham Health Profile | 10 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences Turkey, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Torpil B, Kaya O. Effectiveness of client-centered intervention delivered with face-to-face and telerehabilitation method after total knee arthroplasty-A pilot randomized control trial. Br J Occup Ther. 2022 Jun;85(6):392-399. doi: 10.1177/03080226211070477. Epub 2022 Feb 28. PMID 40336669